CLINICAL TRIAL: NCT03925701
Title: Clinical Study Evaluating the Effectiveness of Vildagliptin Versus Vildagliptin/Metformin on NAFLD With DM
Brief Title: Clinical Study Evaluating Vildagliptin Versus Vildagliptin/Metformin on NAFLD With DM
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sherief Abd-Elsalam (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, Ass. Prof. Tropical Medicine, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: diabetes mellitus tanta
Record Dates: First submitted 2019-04-22; First posted 2019-04-24 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: dm
MeSH Terms: interventions — Vildagliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vildagliptin (Experimental): vildagliptin 50 mg twice daily
  Interventions: Drug: Vildagliptin
- vildagliptin\metformin (Active Comparator): vildagliptin\metformin twice daily
  Interventions: Drug: vildagliptin\metformin

INTERVENTIONS:
Drug: Vildagliptin — vildagliptin twice daily
  Other Names: dibavally
  Arms: vildagliptin
Drug: vildagliptin\metformin — vildagliptin\metformin twice daily
  Other Names: dibavally plus
  Arms: vildagliptin\metformin

SUMMARY:
Clinical study evaluating vildagliptin versus vildagliptin/metformin on NAFLD with DM.

DETAILED DESCRIPTION:
Clinical study evaluating vildagliptin versus vildagliptin/metformin on nonalcoholic fatty liver disease with DM.

ELIGIBILITY:
Inclusion Criteria:

* NAFLD and type 2 DM

Exclusion Criteria:

* Viral hepatitis.
* Child score more than 6.
* renal impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
number of patients with improved nafld and insulin resistance | 6 months
  number of patients showing improved nafld and insulin resistance

CONTACTS AND LOCATIONS:
Overall Officials: Aya G Moussa, Msc, Principal Investigator — Tanta University - Faculty of Pharmacy; Osama M Ibrahim, Prof, Principal Investigator — Prof of Clinical Pharmacy; Gamal Alazab, ass. Prof., Study Director — Prof of Clinical Pharmacy; Yasser Abdel Raouf, Ass Prof, Study Chair — Tanta University-Faculty of Medicine
Locations (1):
- Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No